CLINICAL TRIAL: NCT03933904
Title: A Phase II, Single-arm Open-label Multi-center Study of Sirolimus in Previously Treated Idiopathic Multicentric Castleman Disease
Brief Title: Sirolimus in Previously Treated Idiopathic Multicentric Castleman Disease
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 832465
Record Dates: First submitted 2019-04-29; First posted 2019-05-01 (Actual); Results first posted 2025-08-08 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-07

CONDITIONS: Castleman Disease; Castleman's Disease, Multicentric
Keywords: Castleman; iMCD; Castleman's Disease; multicentric Castleman's disease; multicentric Castleman disease; idiopathic Castleman disease; idiopathic Castleman's disease; CD; MCD; Castleman Disease
MeSH Terms: conditions — Castleman Disease; Multi-centric Castleman's Disease; Macular dystrophy, corneal type 1 | interventions — Sirolimus

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Sirolimus (Experimental): Oral sirolimus: For adults, loading dose of 5 mg/m^2, rounded to the nearest mg, on day 1. For adults, starting on day 2, oral sirolimus daily at 2.5 mg/m^2/day (rounded to the nearest mg), target trough level 10-15 ng/mL by HPLC, for 12 months. For children, 2 mg/m^2/day, target trough level 5-15 ng/mL by HPLC.
  Interventions: Drug: Sirolimus

INTERVENTIONS:
Drug: Sirolimus — Sirolimus (also known as rapamycin) inhibits the mTOR protein kinase and is approved by the USA FDA for the prevention of allograft rejection in renal transplant patients ≥ 13 years of age and for the treatment of lymphangioleiomyomatosis.
  Other Names: Rapamune; Rapamycin

SUMMARY:
The purpose of this study is to understand the impact of sirolimus on idiopathic multicentric Castleman disease.

DETAILED DESCRIPTION:
Human herpesvirus(HHV)-8-negative, idiopathic multicentric Castleman disease (iMCD) is a rare hematologic illness. Current therapeutic options are limited and provide benefit for only a subset of patients. Blockade of IL-6 signaling with siltuximab or tocilizumab abrogates symptoms and improves lymphadenopathy in a portion of patients. However, 66% of patients in the siltuximab Phase II clinical trial did not meet response criteria, and recent studies found that IL-6 is not significantly elevated in many iMCD patients. Recent research has suggested a key role for the phosphoinositide 3-kinase(PI3K)/Akt/mechanistic target of rapamycin (mTOR) pathway in iMCD pathogenesis and off-label administration of sirolimus, an mTOR inhibitor, has shown clinical activity. Based on these experiences, we plan to evaluate the efficacy of sirolimus as a therapy for iMCD patients who are either unable to tolerate anti-IL-6 blockade therapy (siltuximab or tocilizumab), or who fail, relapse, or are refractory to such treatment. This study is a Phase II open label study of daily administration of sirolimus in up to 24 evaluable male or female adults. Participants with iMCD who have failed previous therapy will take daily oral sirolimus for 12 months. Information that is collected as per standard of care will be used to review efficacy, in addition to samples collected specifically for research.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, age 2-80
* Documented disease history consistent with the diagnostic criteria for iMCD
* Failed/refractory (patient did not achieve sufficient disease control with anti-IL-6 therapy, as determined by the site investigator), relapsed (return of symptoms while on therapy), or inability to tolerate anti-IL-6 or anti-IL-6 receptor therapy
* Evidence of active disease, defined as at least two abnormalities in the criteria comprising the CBR criteria, including at least one objective measurement (hemoglobin, weight loss, or lymph node size)
* Ability to consume oral medication in the form of a tablet
* Ability to provide, or for a legally authorized representative to provide on their behalf, informed consent prior to any study-specific activities

Exclusion Criteria:

* Subjects cannot be pregnant or nursing females
* Except for anti-IL6 blockade therapy (siltuximab or tocilizumab), the last dose of which must be ≥ 14 days prior to enrollment (unless subjects cannot or are unwilling to undergo a 14 day washout period), subjects cannot have received any systemic therapy(ies) intended to treat iMCD other than corticosteroids within 28 days of enrollment
* Subjects cannot have previously received sirolimus monotherapy to treat iMCD
* Subjects cannot have any of the following: ECOG >3 (or Karnofsky/Lansky score ≤ 60 in children); Estimated glomerular filtration rate (eGFR) < 30 mL/min/1.73 m2 or creatinine > 3.0 mg/dL; Absolute neutrophil count (ANC) < 1000 x 109/L ((< 500 x 109/L in children); Hemoglobin ≤ 6.5 g/dL (transfusion independent, defined as not receiving a red blood cell transfusion for ≥ 7 days prior); Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) laboratory values greater than three times the upper limit of normal; Albumin < 2 g/dL (transfusion independent, defined as not receiving intravenous albumin for ≥ 7 days prior); Platelet count ≤ 40 x 109/L (transfusion independent, defined as not receiving platelet transfusion for ≥ 7 days prior); Pulmonary involvement or interstitial pneumonitis with dyspnea (adequate pulmonary function is defined as pulse oximetry > 94% on room air if there is clinical indication for determination (e.g. dyspnea at rest, history of interstitial pneumonitis, etc.)); Fasting cholesterol > 300 mg/dL or fasting triglyceride > 400 mg/dL
* Subjects cannot have uncontrolled infection or infectious disease(s) that is/are exclusionary for / mimickers of iMCD
* Subjects cannot have rheumatologic disease(s) that is/are exclusionary for / mimickers of iMCD
* Subjects cannot have a prior malignancy except for: (1) adequately treated basal cell or squamous cell skin cancer, (2) in situ cervical cancer, or (3) other cancer for which the subject has not received treatment within one year prior to enrollment
* Subjects cannot have a documented history of human immunodeficiency virus (HIV) or HHV-8 infection, or severe combined immunodeficiency syndrome
* Subjects cannot have a history of liver or lung transplantation
* Subjects cannot have ongoing or planned participation in another clinical trial involving iMCD directed treatment or that involves immunomodulatory or anti-neoplastic treatment
* Subjects cannot have prior sensitivity / allergy to any formulation of sirolimus, its components or its analogues
* Subjects cannot have serious medical illness, or psychiatric illness or disorders that could potentially interfere with the completion of treatment according to this protocol or participation in the trial
* Subjects cannot have psychiatric disorders that compromises the ability to provide informed consent
* Subjects cannot have any other condition or finding that in the opinion of the investigator would make participation in this trial inappropriate

Ages: 2 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2019-09-25 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2026-06-30 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: David C Fajgenbaum, MD, MBA, MS, Principal Investigator — University of Pennsylvania
Locations (4):
- United States (4):
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - University of California - San Diego, La Jolla, California
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - University of Pennsylvania, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No
There is no current plan to share IPD.

REFERENCES:
- [Derived] van Rhee F, Oksenhendler E, Srkalovic G, Voorhees P, Lim M, Dispenzieri A, Ide M, Parente S, Schey S, Streetly M, Wong R, Wu D, Maillard I, Brandstadter J, Munshi N, Bowne W, Elenitoba-Johnson KS, Fossa A, Lechowicz MJ, Chandrakasan S, Pierson SK, Greenway A, Nasta S, Yoshizaki K, Kurzrock R, Uldrick TS, Casper C, Chadburn A, Fajgenbaum DC. International evidence-based consensus diagnostic and treatment guidelines for unicentric Castleman disease. Blood Adv. 2020 Dec 8;4(23):6039-6050. doi: 10.1182/bloodadvances.2020003334. PMID 33284946
- [Derived] Arenas DJ, Floess K, Kobrin D, Pai RL, Srkalovic MB, Tamakloe MA, Rasheed R, Ziglar J, Khor J, Parente SAT, Pierson SK, Martinez D, Wertheim GB, Kambayashi T, Baur J, Teachey DT, Fajgenbaum DC. Increased mTOR activation in idiopathic multicentric Castleman disease. Blood. 2020 May 7;135(19):1673-1684. doi: 10.1182/blood.2019002792. PMID 32206779
- [Derived] Fajgenbaum DC, Langan RA, Japp AS, Partridge HL, Pierson SK, Singh A, Arenas DJ, Ruth JR, Nabel CS, Stone K, Okumura M, Schwarer A, Jose FF, Hamerschlak N, Wertheim GB, Jordan MB, Cohen AD, Krymskaya V, Rubenstein A, Betts MR, Kambayashi T, van Rhee F, Uldrick TS. Identifying and targeting pathogenic PI3K/AKT/mTOR signaling in IL-6-blockade-refractory idiopathic multicentric Castleman disease. J Clin Invest. 2019 Aug 13;129(10):4451-4463. doi: 10.1172/JCI126091. PMID 31408438

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment started 9/25/2019 and continued until 6/30/2024. Potential participants were informed about the study through various channels, including communication and fliers from licensed site investigators during routine clinical visits. Individuals who previously consented to be contacted for future research were reached by email or phone. Additional outreach was conducted through tools like Epic as well as through the Castleman Disease Collaborative Network (CDCN).
Pre-assignment Details: Before assignment, participants underwent several steps to confirm eligibility. This included a washout period from any systemic therapies used to treat iMCD, as well as various laboratory tests to ensure they were healthy enough to participate and did not have any uncontrolled infections or conditions that could mimic iMCD.
Groups:
- Sirolimus: For adults, the treatment began with a loading dose of 5 mg/m² on Day 1, designed to quickly achieve therapeutic levels of sirolimus. This loading dose was rounded to the nearest milligram and could be adjusted at the discretion of the prescribing physician based on individual tolerability and clinical judgment.
Period: Overall Study
Arm/Group | Sirolimus
Started | 7
Completed | 4
Not Completed | 3

BASELINE CHARACTERISTICS:
Population: 7 patients enrolled into the study with 4 evaluable patients who remained in study for more than 6 weeks.
Groups:
- Sirolimus: Oral sirolimus: Loading dose of 5 mg/m^2, rounded to the nearest mg, on day 1. Starting on day 2, oral sirolimus daily at 2.5 mg/m^2/day (rounded to the nearest mg), target trough level 10-15 ng/mL by HPLC, for 12 months.
Arm/Group | Sirolimus
Number analyzed (Participants) | 7
Age, Continuous [Median (Full Range); unit: years] | 57 [34 to 71]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 7
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 5
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 7
Histopathological Subtype [Count of Participants; unit: Participants]
  Hypervascular/Hyaline Vascular | 1
  Mixed | 3
  Plasmacytic | 1
  Indeterminate | 2
Clinical Subtype [Count of Participants; unit: Participants]
  Thrombocytopenia, Anasarca, Fever, Reticulin fibrosis, and Organomegaly (TAFRO) Subtype | 2
  Idiopathic Plasmacytic Lymphadenopathy (IPL) Subtype | 2
  Not Otherwise Specified (NOS) Subtype | 3

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients Achieving a Positive Clinical Benefit Response (CBR)
Description: Clinical Benefit Response (CBR): The CBR was defined by improvements in clinical symptoms such as fatigue, anorexia, fever, and night sweats.6 Laboratory markers such as hemoglobin levels and weight change were also included in the CBR criteria (Table 1). A CBR was considered positive if there was at least a 25% reduction in the size of the largest lymph node (measured by modified Cheson criteria), a significant improvement in at least one laboratory marker (e.g., hemoglobin), and improvement in at least one clinical symptom without worsening of others.
Time Frame: 12 ± 1 months
Measure: Count of Participants; unit: Participants
Groups:
- Sirolimus: Oral sirolimus: For adults, loading dose of 5 mg/m^2, rounded to the nearest mg, on day 1. For adults, starting on day 2, oral sirolimus daily at 2.5 mg/m^2/day (rounded to the nearest mg), target trough level 10-15 ng/mL by HPLC, for 12 months.
  Sirolimus: Sirolimus (also known as rapamycin) inhibits the mTOR protein kinase and is approved by the USA FDA for the prevention of allograft rejection in renal transplant patients ≥ 13 years of age and for the treatment of lymphangioleiomyomatosis.
Arm/Group | Sirolimus
Number analyzed (Participants) | 4
Participants
  Achieved CBR | 2
  Did Not Achieve CBR | 2

2. Secondary Outcome: Percentage of Patients Achieving a Positive Clinical Benefit Response (CBR) Month 3
Time Frame: Month 3
Measure: Count of Participants; unit: Participants
Arm/Group | Sirolimus
Number analyzed (Participants) | 4
Participants | 1

3. Secondary Outcome: Percentage of Patients Achieving a Positive Clinical Benefit Response (CBR) Month 6
Time Frame: Month 6
Measure: Count of Participants; unit: Participants
Arm/Group | Sirolimus
Number analyzed (Participants) | 4
Participants | 2

4. Secondary Outcome: Percentage of Patients Achieving a Positive Clinical Benefit Response (CBR) Month 9
Time Frame: Month 9
Measure: Count of Participants; unit: Participants
Arm/Group | Sirolimus
Number analyzed (Participants) | 4
Participants | 2

5. Secondary Outcome: Percentage of Patients That Remain on Study Drug for the Duration of the Study
Time Frame: Up to 73 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Sirolimus
Number analyzed (Participants) | 7
Participants | 4

6. Secondary Outcome: Percentage of Patients That Indicate That They Are Currently Receiving Sirolimus at the End of the Follow Up Phase
Time Frame: Up to 73 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Sirolimus
Number analyzed (Participants) | 7
Participants | 1

7. Secondary Outcome: Disease Activity, as Measured by the CHAP Scale
Description: The CHAP scale consists of C-reactive protein (CRP), hemoglobin, albumin, and Eastern Cooperative Oncology Group (ECOG) performance score, each with a subscale range of 0-4. Each criterion in the CHAP scoring system provides a graded measure for a patient's disease activity. The sum of the four scores provides an objective scale for measuring a patient's disease activity and monitoring how it changes over time (scale range 0-16). A higher score indicates greater disease activity.
Time Frame: 12 months ± 2 weeks
Measure: Median (Standard Deviation); unit: score on a scale
Arm/Group | Sirolimus
Number analyzed (Participants) | 4
score on a scale | 3 (0.433)

8. Secondary Outcome: Disease Activity, as Measured by the MCD-related Overall Symptom Score
Description: MCD-related Overall Symptom Score is measured by 34 MCD-related outcome measures. These scores addressed fatigue, weight change, night sweats, etc. The scores were evaluated and graded (as per CTCAE version 4.0, May, 2009), which was used to assess the efficacy of the study intervention. Each symptom score was measured on a numeric scale, ranging from 1 (no symptom) to 5 (very severe or disabling). Scores were combined to create a combined score per patient at each time point. Patients were then assessed as having no response, a symptomatic response, or a durable symptomatic response. A symptomatic response was defined as a ≥50% decrease in the 34-point symptom score, a durable symptomatic response is a ≥50% decrease in the 34-point symptom score from baseline that was maintained for a minimum of 18 weeks.
Time Frame: Month 12
Measure: Count of Participants; unit: Participants
Arm/Group | Sirolimus
Number analyzed (Participants) | 4
Participants
  Achieved a Symptomatic Response | 1
  Achieved a Durable Symptomatic Response | 1
  No Response | 2

9. Secondary Outcome: Proportion of Patients Achieving a Lymph Node Response, Following the Modified Cheson Response Criteria
Description: Radiological response was assessed using the modified Cheson criteria, which quantify changes in lymph node size. A lymph node response was defined as a 25% reduction in bi-dimensional measurements of the largest lymph node compared to baseline. Patients were then assessed according to the following responses:
  Complete Response: All index lesion(s) must have regressed to normal size (≤1.0 cm in their greatest transverse diameter. No new sites of lymphadenopathy >1.5 cm in longest dimension.
  Partial Response: ≥50% decrease in sum of the products of the greatest diameters (SPD) of index lesion(s), and no new sites of lymphadenopathy >1.5 cm in longest dimension.
  Stable Disease: Failure to achieve a CR or PR (see above) without evidence of progressive disease.
  Progressive Disease: ≥50% increase from nadir in the SPD of any index lesion, or appearance of any new sites of lymphadenopathy that measure >1.5 cm in longest dimension during or at the end of therapy.
Time Frame: Month 12
Measure: Number; unit: participants
Arm/Group | Sirolimus
Number analyzed (Participants) | 4
participants
  Achieved Complete Response | 1
  Progressive Disease | 2
  Stable Disease | 1

ADVERSE EVENTS:
Time Frame: Adverse events were collected from baseline to study completion (up to 73 weeks).
Description: Subjects were monitored for all previously reported AEs associated with sirolimus treatment, possible new AEs, and any Grade 2 or higher allergic reaction or hypersensitivity attributed to sirolimus, as judged by the site investigator. AEs were defined according to the NCI CTCAE version 5.0, November 2017. All AEs were recorded in the source document.
Arm/Group | Sirolimus
All-Cause Mortality (participants affected / at risk) | 0/7
Serious Adverse Events (participants affected / at risk) | 1/7
Other Adverse Events (participants affected / at risk) | 7/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sirolimus (N=7)
Pneumonia (Infections and infestations) | 1 (1)
Sepsis (Infections and infestations) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sirolimus (N=7)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (3) — A disorder characterized by an intense itching sensation.
Abdominal pain (Gastrointestinal disorders) | 2 (2)
Bile duct stenosis (Hepatobiliary disorders) | 1 (1)
Blood and lymphatic system disorders-Other, specify (Blood and lymphatic system disorders) | 1 (1) — Neck lymph nodes enlarging
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) — Productive cough
Conjunctivitis (Eye disorders) | 1 (1)
Covid-19 Infection (Infections and infestations) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 2 (2)
Dysphagia (Gastrointestinal disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) — positive d-dimer finding
Eye pain (Eye disorders) | 1 (1)
Headache (Nervous system disorders) | 3 (3)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 2 (2) — Night sweats
Itchy on palms (Skin and subcutaneous tissue disorders) | 1 (1)
Lung infection (Infections and infestations) | 1 (2)
Muscle cramp (Musculoskeletal and connective tissue disorders) | 1 (1) — Cramping of calves and thighs at night
Nausea (Gastrointestinal disorders) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Neuropathy (Nervous system disorders) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (2) — Worsening feet neuropathy; Intermittent numbness and pain in one arm
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Rash acneiform (Skin and subcutaneous tissue disorders) | 1 (2) — hands and head
Shortness of breath (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 1 (1)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Tremors (Nervous system disorders) | 2 (2) — Worsening tremors
Urinary Tract Infection (Infections and infestations) | 1 (1)
Respiratory, thoracic and mediastinal disorders - Other (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Subjective report of being unable to breathe as deeply. Said he has been using albuterol, PRN.
Skin and subcutaneous tissue disorders - Other, specify (ankle) (Skin and subcutaneous tissue disorders) | 1 (1) — Ankle rash
Skin and subcutaneous tissue disorders - Other, specify (groin) (Skin and subcutaneous tissue disorders) | 1 (1)
Skin and subcutaneous tissue disorders - Other, specify (torso) (Skin and subcutaneous tissue disorders) | 1 (1) — Rash on torso
Skin and subcutaneous tissue (Skin and subcutaneous tissue disorders) | 1 (1)
Lump on knee (Musculoskeletal and connective tissue disorders) | 1 (1)
Gastrointestinal disorders - Other (tongue ulcer) (Gastrointestinal disorders) | 1 (1)
Mucositis oral (mouth sores) (Gastrointestinal disorders) | 2 (2)
Generalized muscle weakness (worsening) (Nervous system disorders) | 1 (1)
Fever (General disorders) | 1 (1)
Fatigue (General disorders) | 4 (4) — Stated worst fatigue they've had thus far.
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Dry cough (worsening) (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Chills (General disorders) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Ascites (worsening) (Gastrointestinal disorders) | 2 (2)
Edema limb (leg swelling) (Vascular disorders) | 1 (1)
Lip pain (Gastrointestinal disorders) | 1 (1) — Lips burn
Hypertriglyceridemia (Metabolism and nutrition disorders) | 1 (1)
Swelling of hands and feet (Edema limbs) (Vascular disorders) | 1 (1)
Vascular disorders - Other (Vascular disorders) | 1 (1)
Worsening of night sweats (Skin and subcutaneous tissue disorders) | 1 (1)
Worsening of rash (Skin and subcutaneous tissue disorders) | 1 (1)
Pain (whole body) (Musculoskeletal and connective tissue disorders) | 3 (3) — Intermittent lower leg pain; feeling "achey"

LIMITATIONS AND CAVEATS:
The study's single-arm, open-label design limited conclusions, as there was no control group and potential for bias. The small sample size, impacted by COVID-19 and off-label sirolimus use, reduced statistical power. A short follow-up (12 months plus 12 weeks) limited assessment of long-term efficacy and safety. Given iMCD's chronic nature, future studies should include larger cohorts, control arms, and extended follow-up to assess durability and safety.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-03-20): https://cdn.clinicaltrials.gov/large-docs/04/NCT03933904/Prot_SAP_002.pdf
  • Informed Consent Form (2024-04-11): https://cdn.clinicaltrials.gov/large-docs/04/NCT03933904/ICF_003.pdf